CLINICAL TRIAL: NCT03899649
Title: Registry to Evaluate Effectiveness and Safety of the NanoKnife System for the Ablation of Stage 3 Pancreatic Adenocarcinoma
Brief Title: A Registry Study of NanoKnife IRE for Stage 3 Pancreatic Cancer
Acronym: DIRECT
Status: Active, not recruiting | Type: Observational
Sponsor: Angiodynamics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-ONC-02
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Stage III Pancreatic Cancer
Keywords: Pancreas Cancer; Pancreatic Adenocarcinoma; Pancreatic Ductal Adenocarcinoma; Advanced Pancreatic Cancer; Carcinoma, Pancreatic Ductal; Locally Advanced Pancreatic Cancer; Cancer of Pancreas; Pancreatic Tumor; Pancreatic Carcinoma; Unresectable Pancreatic Cancer; LAPC
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma, Pancreatic Ductal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- IRE Cohort: Patients who received SOC and received IRE
  Interventions: Drug: SOC; Device: NanoKnife System
- SOC Cohort: Patients who received SOC and did not receive IRE
  Interventions: Drug: SOC

INTERVENTIONS:
Drug: SOC — Standard of Care treatment
Device: NanoKnife System — Irreversible Electroporation
  Groups: IRE Cohort

SUMMARY:
This multicenter, observational study will evaluate the effectiveness and safety of the NanoKnife System when used for the ablation of Stage 3 pancreatic adenocarcinoma (Stage 3 PC). Eligible patients will be recruited over a 36-month period and participating institutions will enroll and provide data on consecutive patients that meet inclusion and exclusion criteria. Each patient will be followed up for the duration of the study or until death. The study will include two (2) cohorts: patients who received standard of care (SOC) and received irreversible electroporation (IRE) [IRE cohort], and patients who were treated with SOC and did not receive IRE [SOC cohort].

ELIGIBILITY:
Inclusion Criteria:

1. Provisions of signed and dated informed consent form
2. Patient is 18 years of age and older
3. Patient has a diagnosis of Stage 3 PC cytologically or pathologically confirmed per American Joint Committee on Cancer (AJCC) staging criteria
4. Patient has a tumor evaluated as Stage 3 according to National Comprehensive Cancer Network (NCCN) guidelines, based on radiographic imaging or exploratory surgery
5. Maximum axial and anterior to posterior tumor dimension of ≤3.5cm after SOC
6. Patient has received 3 months of SOC per each participating institution's guidelines
7. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
8. Patient has an American Society of Anesthesiologists (ASA) classification of physical health status of 1 or 2.
9. Patients at IRE sites who are deemed eligible for IRE and receive ablation using the NanoKnife System
10. Patient shows no evidence of disease progression based on NCCN guidelines after completing three (3) months of SOC

Exclusion Criteria:

1. Participation in an interventional trial for pancreatic cancer during the study data collection period
2. Pregnant or lactating patients or male or female patients of reproductive potential who are not willing to employ highly effective birth control from screening to 6 months after the last dose of chemotherapy
3. Patients who are unable to tolerate general anesthetic with full skeletal muscle blockade
4. Patients with the presence of implanted cardiac pacemakers, defibrillators, electronic devices or implanted devices with metal parts in the thoracic cavity at the time of IRE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cytologically or pathologically confirmed Stage 3 PC who are treated, in real-world treatment settings and as part of routine clinical practice, with the NanoKnife System (at least 266 patients) for the ablation of their tumor in addition to SOC (IRE cohort), or with SOC only (at least 266 patients) (SOC cohort). Patients will be enrolled after completing the initial 3-month treatment per SOC for Stage 3 PC.
Sampling Method: Non-Probability Sample
Enrollment: 532 (Estimated)
Dates: Start 2019-05-08 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Time (in months) from time of enrollment to the date of death for any reason, assessed up to 24 months.
  To evaluate the effectiveness of the NanoKnife System when used for the ablation of Stage 3 PC in real world treatment settings, by testing the hypothesis that IRE with the NanoKnife System improves overall survival (OS)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Moores Cancer Center, UC San Diego Health, La Jolla, California
  - University of Florida Health, Gainesville, Florida
  - Miami Cancer Institute, Miami, Florida
  - Wellstar Medical Group, Marietta, Georgia
  - Northwest Community Hospital, Arlington Heights, Illinois
  - University of Iowa Healthcare, Iowa City, Iowa
  - Norton Healthcare, Louisville, Kentucky
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Barnes-Jewish Hospital, St Louis, Missouri
  - NYU Langone, New York, New York
  - Presbyterian Hospital, Columbia, New York, New York
  - Atrium Health, Charlotte, North Carolina
  - St. Luke's University Health Network, Easton, Pennsylvania
  - University of Texas-Southwestern, Dallas, Texas

REFERENCES:
- [Derived] Narayanan G, Bilimoria MM, Hosein PJ, Su Z, Mortimer KM, Martin RCG 2nd. Multicenter randomized controlled trial and registry study to assess the safety and efficacy of the NanoKnife(R) system for the ablation of stage 3 pancreatic adenocarcinoma: overview of study protocols. BMC Cancer. 2021 Jul 7;21(1):785. doi: 10.1186/s12885-021-08474-4. PMID 34233640